CLINICAL TRIAL: NCT05974306
Title: Evaluation of a Proactive Clinical Management and Early Diagnosis of Arrhythmias in Patients With Heart Failure and Non Severely Reduced Left Ventricular Function Through a Telemonitoring System: a Prospective Randomized Clinical Trial (VASCO)
Brief Title: Evaluation of a Proactive Clinical Management and Early Diagnosis of Arrhythmias in Patients With Heart Failure and Non Severely Reduced Left Ventricular Function Through a Telemonitoring System
Acronym: VASCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leonardo Calò, MD (Other)
Responsible Party: Sponsor-Investigator, Leonardo Calò, MD, Principal Investigator, Policlinico Casilino ASL RMB
Organization: Policlinico Casilino ASL RMB (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: v.2.0 29 mar23
Record Dates: First submitted 2023-06-14; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure; Arrhythmias, Cardiac
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILR group (Experimental): patients implanted with an implantable loop recorder to be monitored remotely.
  Interventions: Device: implantable loop recorder
- in-hospital fup group (No Intervention): Patients that will be followed with in-hospital visits.

INTERVENTIONS:
Device: implantable loop recorder — Implantation of an implantable loop recorder
  Arms: ILR group

SUMMARY:
Vasco trial is a no profit, multicenter, international, prospective, randomized study designed to evaluate the clinical benefits of a remote monitoring management based on ILR vs standard practice in patients with high risk of cardiac arrhythmias, heart failure and left ventricle ejection fraction (LVEF)> 40% .The study will enroll about 331 patients (221 in the ILR group and 110 in the in-hospital follow-up group).

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure, LVEF> 40% who report episodes of palpitations.
* Over 18 years of age
* Ability to provide informed consent for registry participation and be willing and able to comply with the protocol described evaluations

Exclusion Criteria:

* Subject who is, or is expected to be unavailable for follow-up
* Pregnancy
* Medical contraindications for ILR implantation
* Patients with PMK / ICD or with Indication for ICD / PMK implantation
* Cardiovascular events / myocardial revascularization in the previous three months
* Patients already on oral anticoagulant treatment
* Patients who do not want to use the telemonitoring system
* Presence of other recognized indications to ILR (Unexplained syncope, cryptogenic stroke/TIA, Transient loss of consciousness and recurrent falls)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the benefits of a remote monitoring management based on ILR vs standard practice in patients with high risk of cardiac arrhythmias, heart failure and LVEF> 40% in the detection of significant clinical events. | 2 years
  Detection rate of arrhythmias that require treatment (medical or interventional)

IPD SHARING:
Plan to Share IPD: No